CLINICAL TRIAL: NCT06059833
Title: Serum Magnesium Level in Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hasnaa Mohamed Kamel, Resident-clinical pathology department-sohag hospital university, Sohag University
Other Study IDs: Soh-Med-23-07-14MS
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases group
  Interventions: Diagnostic Test: Magnesium
- control group
  Interventions: Diagnostic Test: Magnesium

INTERVENTIONS:
Diagnostic Test: Magnesium — The aim of the study is to evaluate serum Mg level in type 2 DM patients.

SUMMARY:
Diabetes mellitus (DM) is a chronic metabolic disorder characterized by persistent hyperglycemia. It may be due to impaired insulin secretion, resistance to peripheral actions of insulin, or both . Chronic hyperglycemia in synergy with the other metabolic aberrations in patients with diabetes mellitus can cause damage to various organ systems, leading to the development of disabling and life-threatening health complications, most prominent of which are microvascular (retinopathy, nephropathy, and neuropathy) and macrovascular complications leading to a 2-fold to 4-fold increased risk of cardiovascular diseases Mg2+ deficiency is usually identified by the measurement of serum Mg2+ concentration. Hypomagnesemia is defined by a serum Mg2+ concentration < 0.75 mmol/L, but a deficiency due to low dietary intake in otherwise healthy people is uncommon. Although overt signs of clinical Mg2+ deficiency are not routinely recognized in the healthy population, relatively low Mg2+ intake and/or Mg2+ status have been shown to be associated with chronic diseases, including cardiovascular disease, T2DM, osteoporosis, pulmonary disease, depression, migraine headaches, inflammation, and cancer

ELIGIBILITY:
Inclusion Criteria:

* • Type 2 Diabetes Mellitus according to WHO criteria.

Exclusion Criteria:

* • Renal failure patients.

  * Type I DM patients.
  * Acute pancreatitis.
  * Hyperthyroidism.
  * Hyperparathyroidism.
  * Malignancies.
  * Patients on loop/thiazide diuretics.
  * Patients on Mg supplement.
  * Patients on Mg containing antacids.
  * Any other conditions causing low Mg levels were excluded from the study.

Min Age: 30 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Type 2 Diabetes Mellitus according to WHO criteria.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
magnesium perecentage | 1 year
  evaluate serum Mg level in type 2 DM patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zheng L, Zhu X, Yang K, Zhu M, Farooqi AA, Kang D, Sun M, Xu Y, Lin X, Feng Y, Liang F, Zhang F, Linhardt RJ. Correction: Zheng, L., et al. PBN11-8, a Cytotoxic Polypeptide Purified from Marine Bacillus, Suppresses Invasion and Migration of Human Hepatocellular Carcinoma Cells by Targeting Focal Adhesion Kinase Pathways. Polymers 2018, 10, 1043. Polymers (Basel). 2021 Jan 5;13(1):166. doi: 10.3390/polym13010166. PMID 33466568
- [Background] Galicia-Garcia U, Benito-Vicente A, Jebari S, Larrea-Sebal A, Siddiqi H, Uribe KB, Ostolaza H, Martin C. Pathophysiology of Type 2 Diabetes Mellitus. Int J Mol Sci. 2020 Aug 30;21(17):6275. doi: 10.3390/ijms21176275. PMID 32872570
- [Background] Piuri G, Zocchi M, Della Porta M, Ficara V, Manoni M, Zuccotti GV, Pinotti L, Maier JA, Cazzola R. Magnesium in Obesity, Metabolic Syndrome, and Type 2 Diabetes. Nutrients. 2021 Jan 22;13(2):320. doi: 10.3390/nu13020320. PMID 33499378
- [Background] Feng J, Wang H, Jing Z, Wang Y, Cheng Y, Wang W, Sun W. Role of Magnesium in Type 2 Diabetes Mellitus. Biol Trace Elem Res. 2020 Jul;196(1):74-85. doi: 10.1007/s12011-019-01922-0. Epub 2019 Nov 11. PMID 31713111